CLINICAL TRIAL: NCT00643565
Title: An Open-label, Multi-center, Randomized Study of the Safety and Effect on Event-free Survival of Bevacizumab in Combination With Standard Chemotherapy in Childhood and Adolescent Patients With Metastatic Rhabdomyosarcoma and Non-rhabdomyosarcoma Soft Tissue Sarcoma
Brief Title: A Study of Avastin (Bevacizumab) in Combination With Standard Chemotherapy in Children and Adolescents With Sarcoma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO20924; 2007-005017-19 (EudraCT Number)
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Bevacizumab

ARMS (2):
- Bevacizumab + Chemotherapy (Experimental): Participants received continuous IV infusion of bevacizumab (7.5 mg/kg every 3 weeks) on Day 1 of 3-week cycles followed by induction chemotherapy (4 cycles of IVADo-containing chemotherapy followed by 5 cycles of IVA-containing chemotherapy) as per institutional practice for a total of 9 cycles during induction treatment phase. As per the investigator decision, local therapy (radiotherapy and /or surgery) was expected to start after 4 weeks of the last bevacizumab administration in the induction phase and resumed to bevacizumab in the maintenance phase at least 4 weeks after the last dose of local therapy. During maintenance treatment phase, participants received IV infusion of bevacizumab (5 mg/kg every 2 weeks) followed by vinorelbine- and cyclophosphamide-containing chemotherapy (as per institutional practice) on Days 1 and 15 of 4-week cycles for a total of 12 cycles.
  Interventions: Drug: Standard chemotherapy; Drug: bevacizumab [Avastin]
- Chemotherapy (Active Comparator): Participants received 9 cycles of induction chemotherapy (4 cycles of IVADo-containing chemotherapy followed by 5 cycles of IVA-containing chemotherapy administered every 3 weeks as per institutional practice. As per the investigator evaluation, participants had option to undergo local therapy (radiotherapy and /or surgery) during last 3 cycles of IVA (i.e. from Cycle 6 to Cycle 9). During maintenance treatment phase, participants received vinorelbine- and cyclophosphamide-containing chemotherapy (as per institutional practice) on Day 1 and 15 of 4-week cycles for a total of 12 cycles.
  Interventions: Drug: Standard chemotherapy

INTERVENTIONS:
Drug: Standard chemotherapy — As prescribed
Drug: bevacizumab [Avastin] — 7.5 mg/kg iv on day 1 of 9 x 3-week cycles, followed by 5 mg/kg iv on days 1 and 15 of each 4-week cycle
  Arms: Bevacizumab + Chemotherapy

SUMMARY:
This open-label two-arm study will assess the safety and efficacy of a combination of bevacizumab + standard chemotherapy with standard chemotherapy alone as active comparator in childhood and adolescent patients with metastatic rhabdomyosarcoma or non-rhabdomyosarcoma soft tissue sarcoma. Patients will be randomized to receive bevacizumab + standard chemotherapy or standard chemotherapy alone. Treatment will consist of 9 x 3-week cycles of induction treatment (standard chemotherapy with or without bevacizumab 7.5 mg/kg iv on day 1 of each cycle) followed by 12 x 4-week cycles of maintenance treatment (standard chemotherapy with or without bevacizumab 5 mg/kg iv on days 1 and 15 of each cycle). The anticipated time on study treatment is 1-2 years.

ELIGIBILITY:
Inclusion Criteria:

* childhood and adolescent patients aged >/=6 months to 18 years of age
* metastatic rhabdomyosarcoma or non-rhabdomyosarcoma soft tissue sarcoma
* adequate bone marrow function
* adequate renal and liver function
* adequate blood clotting

Exclusion Criteria:

* previous malignant tumors
* tumor invading major blood vessels
* prior systemic anti-tumor treatment

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 154 (Actual)
Dates: Start 2008-07-29 (Actual); Primary Completion 2015-05-31 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (61):
- Belgium (3):
  - Hôpital Enfants Reine Fabiola, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Gent, Ghent
- Brazil (6):
  - Instituto Nacional do Cancer - INCA, Rio de Janeiro, Rio de Janeiro
  - Clinica de Oncologia de Porto Alegre - CliniOnco, Porto Alegre, Rio Grande do Sul
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Instituto de Oncologia Pediatrica, São Paulo, São Paulo
  - ITACI - Instituto de Tratamento do Cancer Infantil, São Paulo, São Paulo
  - Hospital Santa Marcelina, São Paulo, São Paulo
- Canada (2):
  - Hospital For Sick Children, Toronto, Ontario
  - Pavillion Chul-Chuq, Sainte-Foy, Quebec
- Hospital Luis Calvo Mackenna; Oncologia, Santiago, Chile
- Czechia (2):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice v Motole, Prague
- France (10):
  - CHU Bordeaux; Unite Onco-Hematologie Pediatrique, Bordeaux
  - Centre Oscar Lambret; Service de Pediatrie, Lille
  - Centre Leon Berard; Pediatrie, Lyon
  - Hopital Timone Enfants; Onco Pediatrie, Marseille
  - Chr De Nantes; Service D'oncologie Pediatrique, Nantes
  - Institut Curie; Oncologie Medicale, Paris
  - CHU Hopital Sud; Service d'Hematologie Pediatrique, Rennes
  - Hopital Des Enfants; Service d Hemato-Oncologie, Toulouse
  - CHU Hopital d Enfants; Centre hospitalier Universitaire Nancy, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy; Service Pediatrique, Villejuif
- Germany (3):
  - University Hospital Essen; Department of Pediatric Oncology, Essen
  - Universitaetsklinikum Freiburg - PS; Partnersite - Onkologie, Freiburg im Breisgau
  - Universitatsklinikum Munster; Padiatrische Hamatologie und Onkologie, Münster
- Israel (4):
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus; Pediatric Hematology Oncology Department, Haifa
  - Schneider Children's Medical Center, Petah Tikva
  - Tel Aviv Sourasky MC, Dana Children's Hospital; Pediatric Hemato-Oncology Clinic, Tel Aviv
- Italy (6):
  - Ospedale Pediatrico Bambino Gesu, Rome, Lazio
  - Istituto Gaslini Ospedale Pediatrico; Dipartimento di Oncoematologia pediatrica, Genoa, Liguria
  - Istituto Nazionale Tumori di Milano; S.C. Oncologia Pediatrica, Milan, Lombardy
  - Dipartimento di Scienze Pediatriche Adolescenza; Osp. Infantile Regina Margherita, Turin, Piedmont
  - U.O.A University Onco-Ematologia Pedicatria; Azienda Ospedaliera A.Meyer, Florence, Tuscany
  - Azienda Ospedaliera di Padova; Clinica di Onco-ematologia pediatrica, Padua, Veneto
- Netherlands (3):
  - Emma Kinderziekenhuis; Dept of Pediatric Oncology, Amsterdam
  - Erasmus Mc/Sophia's Childrens Hospital; Dept. of Pediatric Oncology, Rotterdam
  - Prinses Maxima Centrum, Utrecht
- Poland (2):
  - Uniwersytet Medyczny W Lublinie; Klinika Hematologii i Onkologii Dzieciecej, Lublin
  - Instytut Pomnik-Centrum Zdrowia Dziecka; Klinika Onkologii, Warsaw
- Russia (2):
  - Center for Children's Hematology, Oncology and Immunology, Moscow
  - Saint-Petersburg SHI City Clinical Hospital #31, Saint Petersburg
- Spain (6):
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital Universitari Vall d'Hebron; Servicio de Nefrologia, Barcelona
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital Regional Universitario Carlos Haya;Servicio Oncologia Pediatrica, Málaga
  - Hospital Universitario Virgen del Rocio; Servicio de Onco-Hematologia Pediatrica, Seville
  - Hospital Universitario La Fe, Valencia
- United Kingdom (11):
  - Birmingham Childrens Hospital; Oncology Dept, Birmingham
  - Bristol Royal Hospital For Children, Bristol
  - Royal Hospital for Sick Children, Edinburgh
  - Royal Hospital For Children, Glasgow
  - St. James's University Hospital; Leeds Regional Paediatric Oncology Unit, Leeds
  - Alder Hey Children s Hospital; Department of Pediatrics, Liverpool
  - Great Ormond Street Hospital; Dept. Of Pediatric Oncology, London
  - Royal Manchester Children's Hospital, Manchester
  - The Royal Victoria Infirmary; Paediatric and Adolescent Oncology Unit, Newcastle upon Tyne
  - University Hospital Queens Medical Centre; Department of Paediatric Oncology, Nottingham
  - Royal Marsden Hospital; Pediatric Unit, Surrey

REFERENCES:
- [Derived] Schoot RA, Chisholm JC, Casanova M, Minard-Colin V, Geoerger B, Cameron AL, Coppadoro B, Zanetti I, Orbach D, Kelsey A, Rogers T, Guizani C, Elze M, Ben-Arush M, McHugh K, van Rijn RR, Ferman S, Gallego S, Ferrari A, Jenney M, Bisogno G, Merks JHM. Metastatic Rhabdomyosarcoma: Results of the European Paediatric Soft Tissue Sarcoma Study Group MTS 2008 Study and Pooled Analysis With the Concurrent BERNIE Study. J Clin Oncol. 2022 Nov 10;40(32):3730-3740. doi: 10.1200/JCO.21.02981. Epub 2022 Jun 16. PMID 35709412
- [Derived] Ferrari A, Merks JHM, Chisholm JC, Orbach D, Brennan B, Gallego S, van Noesel MM, McHugh K, van Rijn RR, Gaze MN, Martelli H, Bergeron C, Corradini N, Minard-Colin V, Bisogno G, Geoerger B, Caron HN, De Salvo GL, Casanova M. Outcomes of metastatic non-rhabdomyosarcoma soft tissue sarcomas (NRSTS) treated within the BERNIE study: a randomised, phase II study evaluating the addition of bevacizumab to chemotherapy. Eur J Cancer. 2020 May;130:72-80. doi: 10.1016/j.ejca.2020.01.029. Epub 2020 Mar 13. PMID 32179448
- [Derived] Chisholm JC, Merks JHM, Casanova M, Bisogno G, Orbach D, Gentet JC, Thomassin-Defachelles AS, Chastagner P, Lowis S, Ronghe M, McHugh K, van Rijn RR, Hilton M, Bachir J, Furst-Recktenwald S, Geoerger B, Oberlin O; European paediatric Soft tissue sarcoma Study Group (EpSSG) and the European Innovative Therapies for Children with Cancer (ITCC) Consortium. Open-label, multicentre, randomised, phase II study of the EpSSG and the ITCC evaluating the addition of bevacizumab to chemotherapy in childhood and adolescent patients with metastatic soft tissue sarcoma (the BERNIE study). Eur J Cancer. 2017 Sep;83:177-184. doi: 10.1016/j.ejca.2017.06.015. Epub 2017 Aug 23. PMID 28738258

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chemotherapy | Bevacizumab + Chemotherapy
Started | 80 | 74
Completed | 7 | 7
Not Completed | 73 | 67
Not completed — Death | 12 | 11
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Lost to Follow-up | 0 | 6
Not completed — Other | 7 | 8
Not completed — Refused Treatment / Did Not Cooperate | 0 | 1
Not completed — Recurrence of Disease | 2 | 1
Not completed — Progression of Disease | 18 | 14
Not completed — Protocol Violation | 3 | 0
Not completed — Did Not Cooperate | 0 | 1
Not completed — Administrative | 22 | 16
Not completed — Adverse Event | 5 | 8

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants randomized to the treatment group in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy | Bevacizumab + Chemotherapy | Total
Number analyzed (Participants) | 80 | 74 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.5 (4.8) | 10.3 (4.9) | 10.4 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 29 | 69
  Male | 40 | 45 | 85

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Event-Free Survival (EFS) Events as Per Independent Review Committee (IRC) Assessment
Description: EFS events included tumor progression (IRC assessed), no evidence of response after 3 cycles of induction (derived from IRC assessment), second primary cancer, or death due to any cause. Data for participants who had not experienced an event by the time of clinical cut-off were censored at the date of the last disease assessment prior to the clinical cut-off date. Data for participants who did not have any post-baseline disease assessments were censored at the time of randomization. Tumor progression was defined using Response Evaluation Criteria in Solid Tumors version 1.0 (RECIST v1.0) as at least a 20% increase in the disease measurement, taking as reference the smallest disease measurement recorded since the start of treatment, or the appearance of one or more new lesions, or evidence of clinical progression and unequivocal progression of existing non-target lesions.
Time Frame: Screening up to approximately 6.75 years (assessed at screening, Cycles 4, 7 of induction phase, Cycles 1, 4, 7, 10 of maintenance, then every 3 months for 1.5 years and thereafter every 6 months for 2.5 years)
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 80 | 74
percentage of participants | 52.5 | 68.9

2. Secondary Outcome: Percentage of Participants With Objective Response Prior to First Local Therapy Assessed by RECIST v1.0 Criteria
Description: Objective response prior to first local therapy (surgery and/or radiotherapy) was defined as complete response (CR) or partial response (PR) determined on two consecutive occasions >/=4 weeks apart. Tumor response was assessed as per IRC using RECIST v1.0. CR was defined as disappearance of all target and non-target lesions. If immunocytology was available, no disease was to be detected by that methodology. PR was defined as at least a 30% decrease in the disease measurement, taking as reference the disease measurement done to confirm measurable disease at study entry.
Time Frame: Screening up to approximately 6.75 years
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 80 | 74
percentage of participants | 36.0 [25.23 to 47.91] | 54.0 [40.94 to 66.61]

3. Secondary Outcome: Percentage of Participants Who Experienced EFS Events Among Participants Who Had Objective Response
Description: EFS events was described in Outcome Measure 1 and Outcome Measure 3.
Time Frame: Screening up to approximately 6.75 years
Population: ITT population. Here number of participants analyzed = participants available for the analysis of this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 27 | 34
percentage of participants | 40.7 | 76.5

4. Secondary Outcome: Duration of Response
Description: Duration of Response was defined as time between first objective response and the occurrence of an EFS event (described in Outcome Measure 1). Objective response was defined in Outcome Measure 3. Median duration of response was estimated using Kaplan-Meier estimates and 95% CI for median was computed using the method of Brookmeyer and Crowley.
Time Frame: Screening up to approximately 6.75 years
Population: ITT population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 27 | 34
months | NA [10.18 to NA] — Data was not estimable because of higher number (more than 50%) of censored participants in this arm group. | 17.48 [12.29 to 25.23]

5. Secondary Outcome: Percentage of Participants Who Died
Time Frame: Screening up to approximately 10.75 years (assessed at screening, Cycles 4, 7 of induction phase, Cycles 1, 4, 7, 10 of maintenance, then every 3 months for 1.5 years and thereafter every 6 months for 2.5 years.
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 80 | 74
percentage of participants | 50 | 51.4

6. Primary Outcome: EFS Duration as Per IRC Assessment
Description: EFS was defined as the time between randomization and occurrence of EFS event. EFS events are described in Outcome Measure 1. Median EFS was estimated using Kaplan-Meier estimates and 95% confidence intervals (CI) for median was computed using the method of Brookmeyer and Crowley.
Time Frame: as for outcome 1
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 80 | 74
months | 14.85 [10.84 to 35.88] | 20.63 [15.15 to 24.87]
Statistical Analysis 1: Comparison: Chemotherapy vs Bevacizumab + Chemotherapy; The HR was calculated based on a stratified Cox proportional hazards model, with stratification factors of age and histology/disease risk; Test type: Superiority or Other; p = 0.7189, Log Rank; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.61 to 1.41]

7. Secondary Outcome: Overall Survival Duration
Description: Overall survival was defined as the time between randomization and death due to any cause. Participants without an event were censored at the last time they were known to be alive. Median overall survival was estimated using Kaplan-Meier estimates and 95% CI for median was computed using the method of Brookmeyer and Crowley.
Time Frame: Screening up to approximately 10.75 years (assessed at screening, Cycles 4, 7 of induction phase, Cycles 1, 4, 7, 10 of maintenance, then every 3 months for 1.5 years and thereafter every 6 months for 2.5 years)
Population: ITT population. Here number of participants analyzed = participants available for the analysis of this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 80 | 74
months | 24.02 [17.97 to NA] — Upper limit of 95% CI was not estimable because of the high number (approximately 50%) of censored participants in this arm group | 32.79 [25.33 to NA] — Upper limit of 95% CI was not estimable because of the high number (approximately 50%) of censored participants in this arm group
Statistical Analysis 1: Comparison: Chemotherapy vs Bevacizumab + Chemotherapy; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.3211, Log Rank; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.51 to 1.25]

8. Secondary Outcome: Area Under the Curve at Steady State (AUCss) of Bevacizumab
Description: AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption. AUCss is expressed in milligrams times days per milliliter (mg*day/mL).
Time Frame: Pre- and within 3 hours post-dose on Days 1, 8, and 15 of Cycle 1, Day 1 of Cycle 2-4 of induction phase
Population: Pharmacokinetic (PK)-evaluable population included all randomized participants for whom at least one blood sample was taken for PK assessment following bevacizumab administration. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mg*day/mL
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 70
mg*day/mL | 1010 (256)

9. Secondary Outcome: Volume of Distribution of Bevacizumab
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state.
Time Frame: Pre- and within 3 hours post-dose on Days 1, 8, and 15 of Cycle 1, Day 1 of Cycle 2-4 of induction phase (1 cycle = 3 weeks)
Population: PK-evaluable population. Only participants who received bevacizumab were to be analyzed for PK assessment.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 70
mL | 2070 (891)

10. Secondary Outcome: Half-Life of Bevacizumab
Description: Half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 9
Population: PK-evaluable population. Only participants who received bevacizumab were to be analyzed for PK assessment.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 70
days | 20.8 (8.58)

11. Secondary Outcome: Clearance of Bevacizumab
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body. CL is expressed in milliliters per day (mL/day).
Time Frame: as for outcome 9
Population: PK-evaluable population. Only participants who received bevacizumab were to be analyzed for PK assessment.
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 70
mL/day | 167 (76.4)

ADVERSE EVENTS:
Time Frame: Screening up to approximately 10.75 years.
Description: The safety-evaluable population included all randomized patients who received any dose of study treatment.
Arm/Group | Chemotherapy | Bevacizumab + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 40/79 | 37/71
Serious Adverse Events (participants affected / at risk) | 68/79 | 66/71
Other Adverse Events (participants affected / at risk) | 78/79 | 71/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (N=79) | Bevacizumab + Chemotherapy (N=71)
Anaemia (Blood and lymphatic system disorders) | 3 (8) | 4 (7)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 9 (24) | 19 (49)
Febrile neutropenia (Blood and lymphatic system disorders) | 47 (135) | 46 (120)
Neutropenia (Blood and lymphatic system disorders) | 3 (4) | 2 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiotoxicity (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Fanconi syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Gastrointestinal inflammation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 3 (3) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 4 (5) | 3 (5)
Vomiting (Gastrointestinal disorders) | 7 (8) | 8 (10)
Device related thrombosis (General disorders) | 1 (1) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 7 (14) | 10 (18)
Performance status decreased (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 15 (26) | 14 (14)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Bacteriaemia (Infections and infestations) | 1 (1) | 2 (3)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Candida sepsis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 2 (2) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 3 (3)
Infection (Infections and infestations) | 5 (8) | 3 (6)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic infection (Infections and infestations) | 3 (4) | 4 (7)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Salmonellosis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (4) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Varicella (Infections and infestations) | 0 (0) | 2 (2)
Vulvitis (Infections and infestations) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Recall phenomenon (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Torus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Candida test positive (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (3) | 0 (0)
Neutrophil toxic granulation present (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 3 (3) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (3) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 4 (4)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Vocal cord paresis (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Bladder necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 4 (5) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 1 (1)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Central venous catheter removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Microangiopathy (Vascular disorders) | 0 (0) | 1 (1)
Venoocclusive disease (Vascular disorders) | 1 (1) | 0 (0)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0)
Device Malfunction (Product Issues) | 1 (1) | 0 (0)
Device Dislocation (Product Issues) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy (N=79) | Bevacizumab + Chemotherapy (N=71)
Anaemia (Blood and lymphatic system disorders) | 50 | 55
Febrile neutropenia (Blood and lymphatic system disorders) | 14 | 12
Leukopenia (Blood and lymphatic system disorders) | 11 | 13
Neutropenia (Blood and lymphatic system disorders) | 53 | 56
Thrombocytopenia (Blood and lymphatic system disorders) | 37 | 31
Left ventricular dysfunction (Cardiac disorders) | 4 | 5
Tachycardia (Cardiac disorders) | 4 | 1
Ear pain (Ear and labyrinth disorders) | 4 | 5
Abdominal pain (Gastrointestinal disorders) | 27 | 31
Abdominal pain upper (Gastrointestinal disorders) | 8 | 8
Anal fissure (Gastrointestinal disorders) | 5 | 13
Anal inflammation (Gastrointestinal disorders) | 4 | 6
Constipation (Gastrointestinal disorders) | 40 | 48
Diarrhoea (Gastrointestinal disorders) | 27 | 30
Dyspepsia (Gastrointestinal disorders) | 5 | 4
Mouth ulceration (Gastrointestinal disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 42 | 44
Oral pain (Gastrointestinal disorders) | 4 | 2
Stomatitis (Gastrointestinal disorders) | 23 | 15
Vomiting (Gastrointestinal disorders) | 61 | 64
Asthenia (General disorders) | 10 | 17
Chest pain (General disorders) | 6 | 4
Fatigue (General disorders) | 16 | 18
Mucosal inflammation (General disorders) | 38 | 42
Pain (General disorders) | 10 | 5
Pyrexia (General disorders) | 33 | 27
Hepatocellular injury (Hepatobiliary disorders) | 1 | 4
Hypersensitivity (Immune system disorders) | 1 | 4
Candida infection (Infections and infestations) | 5 | 0
Conjunctivitis (Infections and infestations) | 5 | 7
Ear infection (Infections and infestations) | 3 | 6
Herpes zoster (Infections and infestations) | 4 | 3
Infection (Infections and infestations) | 3 | 5
Nasopharyngitis (Infections and infestations) | 5 | 10
Oral candidiasis (Infections and infestations) | 7 | 5
Paronychia (Infections and infestations) | 0 | 5
Pharyngitis (Infections and infestations) | 0 | 4
Rhinitis (Infections and infestations) | 6 | 12
Upper respiratory tract infection (Infections and infestations) | 7 | 9
Urinary tract infection (Infections and infestations) | 2 | 8
Procedural pain (Injury, poisoning and procedural complications) | 1 | 7
Radiation skin injury (Injury, poisoning and procedural complications) | 12 | 8
Alanine aminotransferase increased (Investigations) | 2 | 6
Gamma-glutamyltransferase increased (Investigations) | 3 | 4
Haemoglobin decreased (Investigations) | 13 | 7
Neutrophil count decreased (Investigations) | 4 | 3
Platelet count decreased (Investigations) | 5 | 4
Weight decreased (Investigations) | 27 | 22
White blood cell count decreased (Investigations) | 2 | 4
Decreased appetite (Metabolism and nutrition disorders) | 18 | 21
Hypokalaemia (Metabolism and nutrition disorders) | 18 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 15
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 | 20
Pain in jaw (Musculoskeletal and connective tissue disorders) | 12 | 5
Dizziness (Nervous system disorders) | 6 | 7
Headache (Nervous system disorders) | 16 | 32
Neuralgia (Nervous system disorders) | 5 | 2
Neuropathy peripheral (Nervous system disorders) | 2 | 9
Paraesthesia (Nervous system disorders) | 3 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 5
Polyneuropathy (Nervous system disorders) | 1 | 4
Anxiety (Psychiatric disorders) | 7 | 9
Insomnia (Psychiatric disorders) | 2 | 5
Dysuria (Renal and urinary disorders) | 3 | 7
Haematuria (Renal and urinary disorders) | 2 | 8
Proteinuria (Renal and urinary disorders) | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 19
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 23
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 22 | 17
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 5
Erythema (Skin and subcutaneous tissue disorders) | 6 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 10
Rash (Skin and subcutaneous tissue disorders) | 10 | 5
Hypotension (Vascular disorders) | 3 | 4
Radiation Injury (Injury, poisoning and procedural complications) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.